CLINICAL TRIAL: NCT03969212
Title: A Phase IIIB, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Clinical Efficacy Study of Baloxavir Marboxil for the Reduction of Direct Transmission of Influenza From Otherwise Healthy Patients to Household Contacts
Brief Title: Study to Assess the Efficacy of Baloxavir Marboxil Versus Placebo to Reduce Onward Transmission of Influenza A or B in Households
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MV40618; 2018-004056-37 (EudraCT Number)
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baloxavir Marboxil (Experimental): Participants who are IPs will receive a single oral dose of baloxavir marboxil. HHCs of the IPs will not receive study medication.
  Interventions: Drug: Baloxavir Marboxil
- Placebo (Placebo Comparator): Participants who are IPs will receive a single oral dose of placebo. HHCs of the IPs will not receive study medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baloxavir Marboxil — IPs less than 12 years old will receive either 2 mg/kg (if weight less than 20 kg) or 40 mg (if weight more than or equal to 20 kg) of Baloxavir Marboxil as oral suspension. IPs more than or equal to 12 years old will receive either 40 mg (if weight less than 80 kg) or 80 mg (if weight more than or equal to 80 kg) of Baloxavir Marboxil as tablets. HHCs of IPs will not receive study medication.
  Other Names: Xofluza
  Arms: Baloxavir Marboxil
Drug: Placebo — IPs less than 12 years old will receive placebo oral suspension and those above 12 years will receive placebo tablets. HHCs of IPs will not receive study medication.
  Arms: Placebo

SUMMARY:
Otherwise healthy index patients (IP) are randomized to either baloxavir marboxil or placebo if their influenza symptoms onset was within 48 hours of screening. Their households are enrolled within 24 hours of randomization if at least 1 household contacts (HHC) have not received influenza vaccine within 6 months of screening and if all HHC screen negative for influenza infection. The main endpoints are assessed based on multiple respiratory swabs, obtained from both IP and HHC up to 9 (+/-1) days post IP randomization, and through the assessment of symptoms.

ELIGIBILITY:
INCLUSION CRITERIA:

Index Patients (IPs):

* Able to comply with the study protocol per investigator judgment.
* Diagnosed with acute influenza infection by investigator.
* Polymerase chain reaction [PCR] (+) or Rapid Influenza Diagnostic Test [RIDT] (+) for influenza A/B based on cobas® SARS-CoV-2 and influenza A/B or other point-of-care / local laboratory results.
* PCR (-) or antigen test (-) for SARS-CoV-2 based on cobas® SARS-CoV-2 and Influenza A/B test or other point-of-care / local laboratory result
* Presence of (a) fever (>=38.0 °C per tympanic or rectal thermometer; >=37.5 °C per axillary, oral or forehead/temporal thermometer) or (b) any influenza symptoms (cough, sore throat, nasal congestion, headache, feverishness or chills, muscle or joint pain, fatigue).
* The time interval between the onset of fever or influenza symptoms and the pre-dose examinations is 48 hours or less.
* IP lives in a household where: (1) No HHC is known to have been diagnosed with influenza or SARS-CoV-2 infection by a healthcare professional (HCP) in the past 4 weeks; (2) All HHCs are expected to meet the key HHC inclusion criteria; (3) >=1 HHCs are expected to participate in the full study who have not received the influenza vaccine within 6 months prior to screening.
* Women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures specified in the protocol

All HHCs (Part 1):

* PCR (-) or RIDT (-) based on cobas® SARS-CoV-2 and influenza A/B or other local point-of-care / local laboratory result.
* PCR (-) or antigen test (-) for SARS-CoV-2 based on cobas® SARS-CoV-2 and Influenza A/B or other POC / local laboratory result.
* HHC lives with no HHC who will be present in the home at any time during the study and who meets any HHC exclusion criteria.
* HHC lives with no HHC who does not meet HHC inclusion criteria (part 1).
* HHC lives in a household where ≥1 HHCs meet all of the following: Start screening within 24 hours after IP randomization; Have NOT received the influenza vaccine within 6 months prior to screening; and Fulfill full study HHC inclusion criteria part 2.

Full study HHCs (part 2) intended for full study must meet the following additional criteria for study entry:

* Agree to participate in the full study.
* Able to comply with the study protocol per investigator judgment
* No influenza symptoms within 7 days prior to screening. Alternatively, mild symptoms are permissible if determined by the investigator to be due to a preexisting condition.
* Temperature <38.0 °C (tympanic).
* Will reside in the index patient's house for at least 7 of the next 9 days and will be present for scheduled study visits.
* Willing and able to measure and record temperature, or have another household member perform the task on his or her behalf. Furthermore, a responsible adult will assume responsibility to oversee or perform this task on behalf of minors.
* In the 6 months prior to screening: a) Has not been diagnosed with influenza by a healthcare professional b) Has not received BXM, peramivir, laninamivir, oseltamivir, zanamivir, rimantadine, umifenovir, favipiravir or amantadine.
* Does not have a moderate or worse active infections OR infections requiring systemic (e.g., oral or intravenous) or otherwise internally administered (e.g., inhaled, intrathecal) antibiotic/antiviral/antifungal therapy, (topical therapies for mild external infections allowed).

EXCLUSION CRITERIA:

IPs:

* IPs with severe influenza virus infection requiring inpatient treatment.
* IPs judged by the investigator to be at high risk for complications of influenza.
* IP is ≥12 years old and unable to swallow tablets (not applicable to IPs 5 to 11 year olds who will receive oral suspension).
* Women who are breastfeeding or have a positive pregnancy test in the pre-dose examinations.
* IPs with concurrent (non-influenza) infections requiring systemic antimicrobial and/or antiviral therapy at the pre-dose examinations.
* IPs who have received baloxavir marboxil, peramivir, laninamivir, oseltamivir, zanamivir, rimantadine, umifenovir, favipiravir or amantadine, or an investigational drug, within 30 days or 5 drug-elimination half-lives, whichever is longer, prior to screening.
* IPs who have received an investigational monoclonal antibody for a viral disease in the last year.
* Known hypersensitivity to baloxavir marboxil or the drug product excipients.
* IP previously included in the study
* IP lives with an HHC who, based on available information, meets the HHC exclusion criteria

HHC:

* Pregnant or within 2 weeks post-partum at screening.
* Immunocompromised.
* Less than 2 years old.
* Who have received an investigational therapy within the 30 days or 5 drug elimination half-lives, whichever is longer, prior to screening.
* Diagnosed with influenza or SARS-CoV-2 infection by a healthcare professional in the past 4 weeks.
* HHC who plans to arrive home after 24 hours post IP randomization to Day 9 and is not willing to be consented as soon as possible upon arrival.
* HHC previously included in the study.

Ages: 5 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4138 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (141):
- United States (42):
  - Cahaba Research, Inc., Birmingham, Alabama
  - Cahaba Research, Inc, Pelham, Alabama
  - Precision Trials, Phoenix, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Long Beach Clinical Trials, Long Beach, California
  - Downtown LA Research Center, Los Angeles, California
  - Probe Clinical Research, Riverside, California
  - MD Strategies Research Centers, San Diego, California
  - Cherry Creek Family Practice, Denver, Colorado
  - Proactive Clinical Research, LLC, Fort Lauderdale, Florida
  - Helios Clinical Research, Inc (former Ventavia Research Group), Kissimmee, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Cordova Research Institute, LLC, Miami, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Kendall South Medical Center Inc., South Miami, Florida
  - Agile Clinical Research Trials, Atlanta, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Mishawaka Osteopathic Clinic, Mishawaka, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Montana Medical Research LLC, Missoula, Montana
  - Accent Clinical Trials, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Hometown Urgent Care and Occupational Health - Springdale, Cincinnati, Ohio
  - Tristar Clinical Investigations, Philadelphia, Pennsylvania
  - Frontier Clinical Research, Scottdale, Pennsylvania
  - Frontier Clinical Research, Smithfield, Pennsylvania
  - Jedda Enterprises dba Galen Clinical Research, Greer, South Carolina
  - AFC Urgent Care-Gunbarrell, Chattanooga, Tennessee
  - Helios Clinical Research, Inc (former Ventavia Research Group), Jackson, Tennessee
  - City Doc Urgent Care-Dallas/Ft. Worth, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Vilo Research Group, Houston, Texas
  - Fairway Medical Clinic, Houston, Texas
  - Mercury Clinical Research, Houston, Texas
  - Family Practice Center, McAllen, Texas
  - Sun Research Institute, San Antonio, Texas
  - Frontier Clinical Research, Kingwood, West Virginia
- Bulgaria (7):
  - Medical Centre "Asklepii", OOD, Dupnitsa
  - Medical Center Hera Eood, Montana
  - MHAT Sveta Paraskeva, Pleven
  - Medizinski Zentrar-1-Sevlievo EOOD, Sevlievo
  - MHAT Sliven - Military Medial Academy, Sliven
  - Medical Center Hera Sofia, Sofia
  - MHAT Sveta Sofia, Sofia
- China (12):
  - Capital Medical University Beijing Hospital of Traditional Chinese Medicine, Beijing
  - Beijing You An Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - The Third People's Hospital of Hainan Province, Sansha
  - Shenzhen People's Hospital, Shenzhen
  - Shenzhen children's hospital, Shenzhen
  - Taizhou People's Hospital, Taizhou
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou
  - General Hospital of Ningxia Medical University, Yinchuan
  - Henan Provincial People's Hospital, Zhengzhou
- ICIMED Instituto de Investigación en Ciencias Médicas, San José, Costa Rica
- Greece (3):
  - Laiko General Hospital - Uni of Athens, Athens
  - Sotiria General Hospital of Athens, Athens
  - Attikon University General Hospital, Chaïdári
- Hungary (4):
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - II. Háziorvosi Körzet, Hosszúhetény
  - Gyermekháziorvosi rendel?- Dr. Újhelyi János, Nyíregyháza
  - OEC Clinical Research, Zalaegerszeg
- JSS Hospital, Mysuru, Karnataka, India
- Israel (2):
  - Kiryat Motzkin Maccabi Medical Center, Kiryat Motzkin
  - Maccabi health services - Moked Hashalom, Tel Aviv
- Japan (43):
  - Toda Internal Medicine & Neurology Clinic, Akashi
  - Medical Corporation Houmankai?Umezu?Clinic, Chikushino-shi
  - Shin Komonji Hospital, Fukuoka
  - Irie Naika Syounika Iin, Fukuoka
  - Kimura Siro Clinic, Fukuoka
  - Iguchi Clinic, Fukuyama
  - Mashiba Clinic, Hannō
  - Fujimaki Ent Clinic, Ichikawa
  - Hisaki Family Clinic, Ichikawa
  - Moriyama Otolaryngology, Kagoshima
  - Kamoike ENT Allergy Clinic, Kagoshima
  - Clinic Kashiwanoha, Kashiwa
  - Kamezawa Clinic, Kasugai
  - Oishi Clinic, Kasuyagun
  - Takahashi naika, Kawasaki
  - Kanagawa Himawari Clinic, Kawasaki
  - Osaki Internal and Respiratory Clinic,, Kitakyushu
  - Morizono medical clinic, Kitakyushu
  - Sato ENT Clinic, Kitakyushu
  - Kiheibashi Otolaryngology, Kodaira
  - Medical corporation Shirayurikai Swing Nozaki Clinic, Musashino
  - Yaesu Clinic, Naha
  - Horikawa Clinic, Nonoichi
  - Lee's Clinic, Osaka
  - Kitada Clinic, Osaka
  - Sunami Internal medicine Clinic, Osaka
  - Funai Ear Nose Throat Clinic, Ōita
  - Saga Memorial Hospital, Saga
  - Segawa Hospital, Saitama
  - Uehara Clinic, Sapporo
  - Aiiku Hospital, Sapporo
  - Tokyo Shinagawa Hospital Medical Corporation Association Tokyokyojuno-kai, Shinagawa City
  - Wakasa Clinic, Tokorozawa
  - Seiwa Clinic, Tokyo
  - Denenchofu Family Clinic, Tokyo
  - Sato Clinic, Tokyo
  - Sekino Hospital, Toshima City
  - Takeru CLINIC, Toyohashi
  - Tsuchiura Beryl Clinic, Tsuchiura
  - Medical corporation Seijinkai Takei Clinic, Tsuru
  - Gushiken-Cardiology and Internal medicine, Urasoe
  - Uranishi Clinic, Urasoe
  - Yotsukaido Tokushukai Medical Center, Yotsukaidō
- Mexico (5):
  - Centro de Investigacion Medico Biologico y Terapia Avanzada, S.C., Guadalajara, Jalisco
  - Centro Respiratorio de México, México, Mexico CITY (federal District)
  - Centro de Estudios Clinicos de Queretaro (CECLIQ), Querétaro City, Querétaro
  - EME RED, Mérida, Yucatán
  - Merida | Investigacion Clinica, Mérida, Yucatán
- Poland (4):
  - KLIMED, Bialystok
  - Centrum Medyczne Lukamed Joanna Luka, Chojnice
  - KO-MED Centra Kliniczne Sp. z o.o., Puławy
  - CLINHOUSE Sp z o.o., Zabrze
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico
- South Africa (4):
  - Into Research, Groenkloof
  - Newtown Clinical Research, Johannesburg
  - Langeberg Clinical Trials, Kraaifontein
  - Midrand Medical Centre, Midrand
- Centro de Salud Las Aguilas, Madrid, Spain
- Turkey (Türkiye) (10):
  - Ankara Bilkent City Hospital, Ankara
  - Ankara University Faculty of Medicine Cebeci Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Atakent Acibadem Private Hosptial Halkali Merkez Mh.,, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Medical Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Karadeniz Technical Uni School of Medicine, Trabzon
- Preston Hill Surgery, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm)

REFERENCES:
- [Derived] Monto AS, Kuhlbusch K, Bernasconi C, Cao B, Cohen HA, Graham E, Hurt AC, Katugampola L, Kamezawa T, Lauring AS, McLean B, Takazono T, Widmer A, Wildum S, Cowling BJ. Efficacy of Baloxavir Treatment in Preventing Transmission of Influenza. N Engl J Med. 2025 Apr 24;392(16):1582-1593. doi: 10.1056/NEJMoa2413156. PMID 40267424
- [Derived] Komeda T, Takazono T, Hosogaya N, Ogura E, Fujiwara M, Miyauchi H, Ajisawa Y, Iwata S, Watanabe H, Honda K, Kitanishi Y, Hara K, Mukae H. Comparison of Household Transmission of Influenza Virus From Index Patients Treated With Baloxavir Marboxil or Neuraminidase Inhibitors: A Health Insurance Claims Database Study. Clin Infect Dis. 2021 Jun 1;72(11):e859-e867. doi: 10.1093/cid/ciaa1622. PMID 33103200

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with acute influenza infection (Index participants [IPs]) and their household contacts (HHCs) took part in the study across 142 investigative sites in 15 countries from 10 October 2019 to 10 May 2024. A total of 4138 participants, 1457 IPs, and 2681 HHCs, were included in the study.
Pre-assignment Details: IPs received baloxavir marboxil or placebo in a 1:1 ratio, and their evaluable HHCs were assessed for influenza symptoms. No treatment was administered to the HHCs. Data was not collected at 'household' level in this study.
Groups:
- Placebo: IPs: IPs were randomized in this arm to receive a single dose of matching placebo orally as a tablet or oral suspension based on their weight and age.
- Baloxavir Marboxil: IPs: IPs were randomized in this arm to receive a single dose of baloxavir marboxil orally based on their weight and age.
- Placebo: HHCs: HHCs related to IPs randomized to the placebo arm were evaluated for influenza transmission (either virological or symptomatic) up to Day 9 of the observation period without any treatment being administered.
- Baloxavir Marboxil: HHCs: HHCs related to IPs randomized to the baloxavir marboxil arm were evaluated for influenza transmission (either virological or symptomatic) up to Day 9 of the observation period without any treatment being administered.
Period: Overall Study
Arm/Group | Placebo: IPs | Baloxavir Marboxil: IPs | Placebo: HHCs | Baloxavir Marboxil: HHCs
Started | 731 | 726 | 1336 | 1345
Treated (Safety IP Set included all randomized participants who received at least one dose of study treatment. One participant was randomized to placebo but received baloxavir and is counted in the Baloxavir arm for safety analysis.) | 726 (Treated with Placebo.) | 723 (Treated with Baloxavir Marboxil.) | 0 | 0
Completed | 699 | 688 | 1300 | 1305
Not Completed | 32 | 38 | 36 | 40
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 13 | 5 | 11
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Reason not Specified | 22 | 23 | 28 | 26

BASELINE CHARACTERISTICS:
Population: Full Index Participant Analysis Set (FAS-IP) included all randomized IPs. Full Household Contact Analysis Set (FAS-HC) included all HHCs who were enrolled for the full study and linked to a randomized IP, regardless of polymerase chain reaction (PCR) test status of IP for influenza A or B. Baseline data was not collected for four participants from the 'Baloxavir Marboxil: HHCs' arm, hence data for 1341 participants is presented here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo: IPs | Baloxavir Marboxil: IPs | Placebo: HHCs | Baloxavir Marboxil: HHCs | Total
Number analyzed (Participants) | 731 | 726 | 1336 | 1341 | 4134
Age, Customized [Count of Participants; unit: Participants]
  2-11 years | 65 | 65 | 152 | 151 | 433
  12-17 years | 120 | 118 | 133 | 124 | 495
  18-64 years | 546 | 543 | 985 | 989 | 3063
  65-84 years | 0 | 0 | 61 | 71 | 132
  ≥ 85 years | 0 | 0 | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 377 | 389 | 740 | 709 | 2215
  Male | 354 | 337 | 596 | 632 | 1919
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 83 | 169 | 153 | 488
  Not Hispanic or Latino | 646 | 633 | 1133 | 1145 | 3557
  Unknown or Not Reported | 2 | 10 | 34 | 43 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 7 | 9 | 8 | 31
  Asian | 196 | 190 | 370 | 364 | 1120
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 10 | 0 | 10
  Black or African American | 28 | 19 | 47 | 46 | 140
  White | 483 | 495 | 817 | 871 | 2666
  More than one race | 3 | 0 | 9 | 5 | 17
  Unknown or Not Reported | 14 | 15 | 74 | 47 | 150

OUTCOME MEASURES:

1. Primary Outcome: Percentage of HHCs With Virological Influenza Transmission by Day 5
Description: The virological transmission was determined based on Polymerase Chain Reaction Positive (PCR+) influenza test results. The adjusted incidence (cumulative proportion of events by Day 5) rate is reported here. This is defined as percentage of HHCs who tested PCR+ for influenza by Day 5 post IP randomization with virus subtype matching with that of the respective IP, irrespective of being symptomatic or asymptomatic. The adjusted incidence rates presented were estimated using a generalized estimating equations (GEE) approach.
Time Frame: Baseline (Day 1) to Day 5
Population: The primary household contacts analysis set (PAS-HC) included unvaccinated HHCs who were linked to households where the IP was baseline PCR+ for influenza A or B, received the study drug, and where all contacts were PCR negative at baseline.
Measure: Number (95.38% Confidence Interval); unit: percentage of HHCs
Arm/Group | Placebo: HHCs | Baloxavir Marboxil: HHCs
Number analyzed (Participants) | 1098 | 1118
percentage of HHCs | 13.42 [10.66 to 16.76] | 9.50 [7.40 to 12.13]
Statistical Analysis 1: Comparison: Placebo: HHCs vs Baloxavir Marboxil: HHCs; The odds ratio (OR) shown represents the odds of Baloxavir Marboxil (BMX) versus the odds of Placebo; Test type: Superiority; p = 0.013, GEE; Adjusted OR (BMX vs Placebo) = 0.68, 95.38% CI 2-sided [0.50 to 0.93]

2. Secondary Outcome: Percentage of HHCs With Symptomatic Influenza Transmission by Day 5
Description: The adjusted incidence (cumulative proportion of events by Day 5) rate is reported here. This is defined as percentage of HHCs who tested PCR+ for influenza by Day 5 post IP randomization with virus subtype matching with that of respective IP, & developed symptoms at any time during the study. The adjusted incidence rates presented were estimated using a GEE approach. HHCs ≥12 years old were symptomatic if 1. Presence of temperature ≥38.0 Celsius (C) and 1 respiratory symptom (cough, sore throat, nasal congestion) or 2. Presence of 1 respiratory symptom and 1 general systemic symptom (headache, feverishness or chills, muscle or joint pain, fatigue), with/without a fever. HHCs ≥2 and <12 years old were symptomatic if the presence of temperature was ≥38.0°C and had upper respiratory tract infection signs or symptoms (cough, nasal congestion, or rhinorrhea). Symptoms must be either new or have worsened versus baseline in HHC with baseline symptoms due to a preexisting comorbidity.
Time Frame: Baseline (Day 1) to Day 5
Population: PAS-HC included unvaccinated HHCs who were linked to households where the IP was baseline PCR+ for influenza A or B, received the study drug, and where all contacts were PCR negative at baseline.
Measure: Number (95.38% Confidence Interval); unit: percentage of HHCs
Arm/Group | Placebo: HHCs | Baloxavir Marboxil: HHCs
Number analyzed (Participants) | 1098 | 1118
percentage of HHCs | 7.61 (5.66) [5.66 to 10.17] | 5.80 (4.10) [4.10 to 8.15]
Statistical Analysis 1: Comparison: Placebo: HHCs vs Baloxavir Marboxil: HHCs; The OR shown represents the odds of BMX versus the odds of Placebo; Test type: Superiority; p = 0.1550, GEE model; Adjusted OR (BMX vs Placebo) = 0.75, 95.38% CI 2-sided [0.50 to 1.12]

3. Secondary Outcome: Percentage of Households (HHs) With Virological Influenza Transmission at Household Level by Day 5
Description: Percentage of households with at least one HHC who met the primary endpoint of virological transmission by Day 5 are reported here. 'Number of participants analyzed' is the number of IPs in the PAS-IP set.
Time Frame: Baseline (Day 1) to Day 5
Population: Primary Households Analysis Set (PAS-HH) included all households of randomized IPs that were PCR+ at screening and with at least one HHC enrolled for the full study. IPs should be a part of the Primary Index Patients Analysis Set (PAS-IP) which includes all randomized IPs with at least 1 HHC in the PAS-HC. PAS-HC included unvaccinated HHCs who were linked to households where the IP was baseline PCR+ for influenza A/B, received study drug, and where all contacts were PCR negative at baseline.
Measure: Number; unit: percentage of HHs
Units Other Than Participants: Households
Groups:
- Placebo: IPs: IPs were randomized in this arm to receive a single dose of matching placebo orally as a tablet or oral suspension based on their weight and age.
  All households of randomized IPs who received matching placebo, with the IP being PCR positive at screening and with at least one HHC enrolled for the full study were assessed.
- Baloxavir Marboxil: IPs: IPs were randomized in this arm to receive a single dose of baloxavir marboxil orally based on their weight and age.
  All households of randomized IPs who received baloxavir marboxil, with the IP being PCR positive at screening and with at least one HHC enrolled for the full study were assessed.
Arm/Group | Placebo: IPs | Baloxavir Marboxil: IPs
Number analyzed (Participants) | 544 | 548
Number analyzed (Households) | 544 | 548
percentage of HHs | 19.5 | 15.5
Statistical Analysis 1: Comparison: Placebo: IPs vs Baloxavir Marboxil: IPs; The OR shown represents the odds of BMX versus the odds of Placebo; Test type: Other; Odds Ratio (BMX vs Placebo}] = 0.76, 95.38% CI 2-sided [0.55 to 1.06]

4. Secondary Outcome: Percentage of HHs With Symptomatic Influenza Transmission at Household Level by Day 5
Description: Percentage of HHs with at least one HHC who meets the symptomatic transmission by Day 5 endpoint are reported here. 'Number of participants analyzed' is the number of IPs in the PAS-IP set.
Time Frame: Baseline (Day 1) to Day 5
Population: PAS-HH included all households of randomized IPs that were PCR+ at screening and with at least one HHC enrolled for the full study. The IPs should be a part of the PAS-IP which includes all randomized IPs with at least one HHC in the PAS-HC. PAS-HC included unvaccinated HHCs who were linked to households where the IP was baseline PCR+ for influenza A or B, received the study drug, and where all contacts were PCR negative at baseline.
Measure: Number; unit: percentage of HHs
Units Other Than Participants: Households
Arm/Group | Placebo: IPs | Baloxavir Marboxil: IPs
Number analyzed (Participants) | 544 | 548
Number analyzed (Households) | 544 | 548
percentage of HHs | 11.9 | 8.6
Statistical Analysis 1: Comparison: Placebo: IPs vs Baloxavir Marboxil: IPs; The OR shown represents the odds of BMX versus the odds of Placebo; Test type: Other; Odds Ratio (BMX vs Placebo) = 0.69, 95.38% CI 2-sided [0.46 to 1.04]

5. Secondary Outcome: Percentage of HHCs With Virological Influenza Transmission by Day 9
Description: The adjusted incidence (cumulative proportion of events by Day 9) rate is reported here. This is defined as percentage of HHCs who tested PCR+ for influenza by Day 9 post IP randomization with virus subtype matching with the respective IP, irrespective of being symptomatic or asymptomatic including: 1. all HHC meeting primary endpoint, AND 2. all HHC cases detected after Day 5 meeting the following criteria: 2a. included HHC case was in an HH where another HHC had already met the primary endpoint OR 2b. included HHC case was PCR+ bearing an amino acid substitution of isoleucine for another amino acid at position 38 (I38X) in the polymerase acidic (PA) protein (PA/I38X substitution) or amino acid substitution of threonine to lysine at position 20 in the PA protein for influenza B only (PA/T20K). The adjusted incidence rates presented were estimated using a GEE approach.
Time Frame: Baseline (Day 1) to Day 9
Population: PAS-HC analysis set included unvaccinated HHCs who were linked to households where the IP was baseline PCR+ for influenza A or B, received the study drug, and where all contacts were PCR negative at baseline. Overall number analyzed included number of HHCs with data available for analysis.
Measure: Number (95.38% Confidence Interval); unit: percentage of HHCs
Arm/Group | Placebo: HHCs | Baloxavir Marboxil: HHCs
Number analyzed (Participants) | 1038 | 1081
percentage of HHCs | 15.40 (12.20) [12.20 to 19.27] | 10.77 (8.41) [8.41 to 13.71]
Statistical Analysis 1: Comparison: Placebo: HHCs vs Baloxavir Marboxil: HHCs; The OR shown represents the odds of BMX versus the odds of Placebo; Test type: Other; GEE model; Adjusted OR (BMX vs Placebo) = 0.66, 95.38% CI 2-sided [0.48 to 0.91]

6. Secondary Outcome: Percentage of HHCs With Symptomatic Influenza Transmission by Day 9
Description: The adjusted incidence (cumulative proportion of events by Day 9) rate is reported here. This is defined as percentage of HHCs who met the virological transmission by Day 9 endpoint and developed symptoms at any time during the study. The adjusted incidence rates presented were estimated using a GEE approach. HHCs ≥12 years were symptomatic if they had 1. temperature ≥38.0°C and one respiratory symptom (cough, sore throat, nasal congestion) or 2. one respiratory and one general systemic symptom (headache, feverishness or chills, muscle or joint pain, fatigue), with or without fever. HHCs ≥2 and <12 years were symptomatic if the presence of temperature was ≥38.0°C and had upper respiratory symptoms (headache, feverishness or chills, muscle or joint pain, fatigue). Symptoms must be either new or have worsened versus baseline in HHC with baseline symptoms due to a preexisting comorbidity.
Time Frame: Baseline (Day 1) to Day 9
Population: PAS-HC included unvaccinated HHCs who were linked to households where IP was baseline PCR+ for influenza A or B, received study drug, and where all contacts were PCR negative at baseline. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number (95.38% Confidence Interval); unit: percentage of HHCs
Arm/Group | Placebo: HHCs | Baloxavir Marboxil: HHCs
Number analyzed (Participants) | 1037 | 1079
percentage of HHCs | 8.26 [6.10 to 11.09] | 6.15 [4.37 to 8.58]
Statistical Analysis 1: Comparison: Placebo: HHCs vs Baloxavir Marboxil: HHCs; The OR shown represents the odds of BMX versus the odds of Placebo; Test type: Other; Two-Sided P-value; Adjusted OR (BMX vs Placebo) = 0.73, 95.38% CI 2-sided [0.48 to 1.09]

7. Secondary Outcome: Percentage of HHCs With Any Virological Infection by Day 9
Description: Virological infection was defined as HHCs who tested PCR+ for influenza by Day 9 post IP randomization based on PCR influenza test results. The adjusted incidence (cumulative proportion of events by Day 9) rate is reported here. This is defined as percentage of HHCs who met the virological infection by Day 9 endpoint. The adjusted incidence rates presented were estimated using a GEE approach.
Time Frame: Baseline (Day 1) to Day 9
Population: PAS-HC included unvaccinated HHCs who were linked to households where the IP was baseline PCR+ for influenza A or B and received study drug and where all contacts were PCR negative at baseline. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number (95.38% Confidence Interval); unit: percentage of HHCs
Arm/Group | Placebo: HHCs | Baloxavir Marboxil: HHCs
Number analyzed (Participants) | 1040 | 1071
percentage of HHCs | 18.68 (15.36) [15.36 to 22.53] | 13.98 (11.31) [11.31 to 17.16]
Statistical Analysis 1: Comparison: Placebo: HHCs vs Baloxavir Marboxil: HHCs; The OR shown represents the odds of BMX versus the odds of Placebo; Test type: Other; Two-Sided P-value; Adjusted OR (BMX vs Placebo) = 0.71, 95.38% CI 2-sided [0.53 to 0.94]

8. Secondary Outcome: Percentage of HHs With Any Virological Infection at HH Level by Day 9
Description: Virological infection at the HH level was defined as the HHs with at least one HHC who met the endpoint of any virological infection by Day 9. 'Number of participants analyzed' is the number of IPs in the PAS-IP set.
Time Frame: Baseline (Day 1) to Day 9
Population: as for outcome 4
Measure: Number; unit: percentage of HHs
Units Other Than Participants: Households
Arm/Group | Placebo: IPs | Baloxavir Marboxil: IPs
Number analyzed (Participants) | 544 | 548
Number analyzed (Households) | 544 | 548
percentage of HHs | 24.3 | 20.1
Statistical Analysis 1: Comparison: Placebo: IPs vs Baloxavir Marboxil: IPs; The OR shown represents the odds of BMX versus the odds of Placebo; Test type: Other; Odds Ratio (BMX vs Placebo) = 0.79, 95.38% CI 2-sided [0.59 to 1.06]

9. Secondary Outcome: Percentage of HHCs With Any Symptomatic Infection by Day 9
Description: The adjusted incidence (cumulative proportion of events by Day 9) rate is reported here. This is defined as percentage of HHCs who tested PCR+ for influenza by Day 9 post IP randomization and developed symptoms at any time during the study. The adjusted incidence rates presented were estimated using a GEE approach. HHCs ≥12 years were symptomatic if they had (1) a temperature ≥38.0°C and one respiratory symptom (cough, sore throat, nasal congestion) or (2) one respiratory and one systemic symptom (headache, chills, muscle/joint pain, fatigue), with or without fever. HHCs ≥2 and <12 years were symptomatic if the presence of temperature was ≥38.0°C and had upper respiratory symptoms (cough, nasal congestion, rhinorrhea). Symptoms must be either new or have worsened versus baseline in HHC with baseline symptoms due to a preexisting comorbidity.
Time Frame: Baseline (Day 1) to Day 9
Population: as for outcome 7
Measure: Number (95.38% Confidence Interval); unit: percentage of HHCs
Arm/Group | Placebo: HHCs | Baloxavir Marboxil: HHCs
Number analyzed (Participants) | 1039 | 1069
percentage of HHCs | 8.71 (6.49) [6.49 to 11.60] | 6.43 (4.61) [4.61 to 8.91]
Statistical Analysis 1: Comparison: Placebo: HHCs vs Baloxavir Marboxil: HHCs; The OR shown represents the odds of BMX versus the odds of Placebo; Test type: Other; Two-Sided P-value; Adjusted OR (BMX vs Placebo) = 0.72, 95.38% CI 2-sided [0.49 to 1.07]

10. Secondary Outcome: Percentage of HHs With Any Symptomatic Infection at HH Level by Day 9
Description: Percentage of HHs with at least one HHC who meets the endpoint of any symptomatic infection by Day 9 are reported here. HHCs ≥12 years were symptomatic if they had 1. a temperature ≥38.0°C &1 respiratory symptom (cough, sore throat, nasal congestion) or 2. 1 respiratory & 1 systemic symptom (headache, chills, muscle/joint pain, fatigue), with/without fever. HHCs ≥2 & <12 years were symptomatic if the temperature was ≥38.0°C & had upper respiratory symptoms (cough, nasal congestion, rhinorrhea). Symptoms must be new or have worsened versus baseline in HHC with baseline symptoms due to preexisting comorbidity. 'Number of participants analyzed' is the number of IPs in the PAS-IP set.
Time Frame: Baseline (Day 1) to Day 9
Population: as for outcome 4
Measure: Number; unit: percentage of HHs
Units Other Than Participants: Households
Arm/Group | Placebo: IPs | Baloxavir Marboxil: IPs
Number analyzed (Participants) | 544 | 548
Number analyzed (Households) | 544 | 548
percentage of HHs | 12.9 | 9.5
Statistical Analysis 1: Comparison: Placebo: IPs vs Baloxavir Marboxil: IPs; The OR shown represents the odds of BMX versus the odds of Placebo; Test type: Other; Odds Ratio (BMX vs Placebo) = 0.71, 95.38% CI 2-sided [0.48 to 1.04]

11. Secondary Outcome: Number of IPs With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: Baseline up to Day 9 (for IPs ≥12 years old) and Day 21 (for IPs <12 years old)
Population: Safety IP Set included all randomized participants who received at least one dose of study treatment. One participant was randomized to placebo but received baloxavir and is counted in the Baloxavir arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: IPs | Baloxavir Marboxil: IPs
Number analyzed (Participants) | 726 | 723
Participants | 51 | 33

12. Secondary Outcome: Number of IPs With Serious Adverse Events (SAEs)
Description: A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Baseline up to Day 9 (for IPs ≥12 years old) and Day 21 (for IPs <12 years old)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: IPs | Baloxavir Marboxil: IPs
Number analyzed (Participants) | 726 | 723
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Day 9 (IPs ≥12 years old) Baseline up to Day 21 (IPs <12 years old)
Description: Safety IP Set included all randomized participants who received at least one dose of study treatment. One participant was randomized to placebo but received baloxavir and is counted in the Baloxavir arm. Safety data was collected only for IPs as no treatment was administered to the HHCs in this study.
Groups:
- Baloxavir Marboxil: IPs: IPs received a single dose of baloxavir marboxil orally based on their weight and age.
Arm/Group | Placebo: IPs | Baloxavir Marboxil: IPs
All-Cause Mortality (participants affected / at risk) | 0/726 | 0/723
Serious Adverse Events (participants affected / at risk) | 2/726 | 1/723
Other Adverse Events (participants affected / at risk) | 0/726 | 0/723
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: IPs (N=726) | Baloxavir Marboxil: IPs (N=723)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT03969212/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03969212/SAP_001.pdf